CLINICAL TRIAL: NCT02542553
Title: Bilateral Bronchoalveolar Lavage Cultures for Diagnosing Ventilator-associated Pneumonia. Microbiologic Concordance and Impact on the Efficacy of Treatment Decisions.
Brief Title: Bilateral Bronchoalveolar Lavage in Ventilator-associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giuseppe Bello, Medical doctor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Bilateral BAL in VAP
Record Dates: First submitted 2015-08-25; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bilateral BAL (Experimental): Bronchoscopies are performed in strict accordance with consensus guidelines. The left or right lung is examined with a flexible fiberoptic bronchoscope. If localized infiltrates are present on the chest radiograph, the tip of the scope is wedged into a subsegment of the area displaying the most marked opacity. In the presence of diffuse opacity or when no clear roentgenographic abnormalities are observed, the tip is positioned in the lingula or right middle lobe. Five 20-ml aliquots of sterile normal saline are then injected and reaspirated with a syringe. Bronchoscopy is then repeated in the same manner in the contralateral lung with a second, sterile bronchoscope of the same brand and model.
  Interventions: Procedure: Bilateral BAL

INTERVENTIONS:
Procedure: Bilateral BAL

SUMMARY:
The purpose of this study is to assess microbiologic concordance rates between right- and left-lung bronchoalveolar lavage cultures from patients with suspected ventilator-associated pneumonia, identify predictors of concordance, and evaluate the impact of discordant microbiology on clinicians' ability to prescribe appropriate antibiotic treatments, the investigators conducted a prospective observational study in the general intensive care unit of a large university hospital.

DETAILED DESCRIPTION:
Bronchoscopic sampling of lower respiratory tract secretions is widely used in intensive care units (ICUs) for the microbiological diagnosis of ventilator-associated pneumonia (VAP). However, the importance of selecting a specific lung segment for sampling is still a matter of debate.

Non-bronchoscopic blind mini-bronchoalveolar lavage (BAL) is currently used for the diagnosis of VAP with satisfactory sensitivity and specificity. In the presence of pneumonia, microbiologic concordance between the left and right lungs becomes crucial. If concordance is low, the reliability of blind sampling becomes questionable.

When the bacterial distribution in the right and left lungs of VAP patients has been investigated using bronchoscopic sampling techniques, rates of microbiological concordance between the two specimens have varied widely (from 53% to 92%). The factors potentially associated with concordant culture yields have never been explored, and it is unclear whether the use of guided, bilateral lung sampling would actually improve the appropriateness of the antibiotic regimens prescribed for patients with suspected VAP.

The primary objective of this study is to assess the frequency of microbiologic concordance between the right- and left-lung samples in ICU patients undergoing bronchoscopic BAL performed with two different fiberoptic bronchoscopes for the suspicion of VAP. Secondary objectives are to identify factors associated with such concordance and to evaluate the suitability of treatments prescribed based on unilateral vs. bilateral BAL cultures.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation of ≥ 48 hours
* clinically suspected pneumonia (simplified Clinical Pulmonary Infectious Score exceeded 6 or chest radiographs with a new or progressive pulmonary infiltrate in a patient with at least two of the following: purulent respiratory secretions, temperature >38°C or <36°C, white blood cell count >12,000/mm3 or <4,000/mm3)

Exclusion Criteria:

* age <18 years
* pregnancy
* absence of informed consent
* an arterial oxygen partial pressure to inspired oxygen fraction ratio (PaO2:FiO2) of ≤150
* use of positive end-expiratory pressure (PEEP) >10 cmH2O
* active uncontrolled bronchospasm
* unstable angina or recent (<6 weeks) myocardial infarction
* unstable arrhythmia
* intracranial hypertension
* platelet count ≤20,000/mm3
* international normalized ratio (INR) or activated partial thromboplastin time (aPTT) ratio >1.5
* documented treatment-limitation orders in the patient's chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Rate of microbiologic concordance between the right- and left-lung samples | After at least 48 hours of invasive mechanical ventilation
  Pneumonia is microbiologically confirmed when the quantitative culture of one or both BAL specimens is positive at significant growth for at least one potential bacterial pathogen. Right and left BAL cultures are classified as concordant when both are positive for the same organism(s) or when neither show any growth. Cultures are classified as discordant when at least one of the microorganisms isolated from one specimen is not recovered from the contralateral specimen.

SECONDARY OUTCOMES:
Possible association between purulent secretions and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between duration of mechanical ventilation and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between duration of ICU stay and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between duration of hospital stay and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between immunosuppression and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between antibiotic treatment and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between radiological infiltrate and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between body temperature and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between WBC count and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between PaO2:FiO2 and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between PEEP and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between CPIS and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between type of humidification and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between procalcitonin and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy
Possible association between C-reactive protein and microbiologic concordance between right- and left-lung BAL cultures | At an expected average of 48 hours after bronchoscopy

OTHER OUTCOMES:
Comparison of antibiotic regimens chosen on the basis of right or left-lung culture results alone with regimens chosen on the basis of bilateral culture results, by performing a simulated prescribing experiment. | At 18 months after study initiation
  For each enrolled patient, actual treatment decisions are made by the ICU attending physicians in charge of the case on the basis of the results of bilateral BAL culture and sensitivity analyses. Later, at the end of the study, data for patients with discordant BAL cultures are reviewed in a simulated prescribing session by a second team composed of an ICU physician and an infectious disease specialist. The team is asked to propose an appropriate antimicrobial regimen based on the culture and in vitro antimicrobial susceptibility data for the right-lung BAL sample alone, the left-lung BAL sample alone, and the right and left BAL samples. Each microbiological report is presented separately to the team with a summary of the patient's relevant clinical data. The prescribed regimen is defined as appropriate if it provides active coverage for all of the organisms identified in both BAL specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Bello, MD, Principal Investigator — Università Cattolica del Sacro Cuore, Rome, Italy

REFERENCES:
- [Result] Meduri GU, Chastre J. The standardization of bronchoscopic techniques for ventilator-associated pneumonia. Chest. 1992 Nov;102(5 Suppl 1):557S-564S. doi: 10.1378/chest.102.5_supplement_1.557s. No abstract available. PMID 1424930
- [Result] Marquette CH, Herengt F, Saulnier F, Nevierre R, Mathieu D, Courcol R, Ramon P. Protected specimen brush in the assessment of ventilator-associated pneumonia. Selection of a certain lung segment for bronchoscopic sampling is unnecessary. Chest. 1993 Jan;103(1):243-7. doi: 10.1378/chest.103.1.243. PMID 8417887
- [Result] Meduri GU, Reddy RC, Stanley T, El-Zeky F. Pneumonia in acute respiratory distress syndrome. A prospective evaluation of bilateral bronchoscopic sampling. Am J Respir Crit Care Med. 1998 Sep;158(3):870-5. doi: 10.1164/ajrccm.158.3.9706112. PMID 9731019
- [Result] Butler KL, Best IM, Oster RA, Katon-Benitez I, Lynn Weaver W, Bumpers HL. Is bilateral protected specimen brush sampling necessary for the accurate diagnosis of ventilator-associated pneumonia? J Trauma. 2004 Aug;57(2):316-22. doi: 10.1097/01.ta.0000088858.22080.cb. PMID 15345979
- [Result] Jackson SR, Ernst NE, Mueller EW, Butler KL. Utility of bilateral bronchoalveolar lavage for the diagnosis of ventilator-associated pneumonia in critically ill surgical patients. Am J Surg. 2008 Feb;195(2):159-63. doi: 10.1016/j.amjsurg.2007.09.030. PMID 18096127
- [Result] Zaccard CR, Schell RF, Spiegel CA. Efficacy of bilateral bronchoalveolar lavage for diagnosis of ventilator-associated pneumonia. J Clin Microbiol. 2009 Sep;47(9):2918-24. doi: 10.1128/JCM.00747-09. Epub 2009 Jul 15. PMID 19605577
- [Result] Esperatti M, Ferrer M, Theessen A, Liapikou A, Valencia M, Saucedo LM, Zavala E, Welte T, Torres A. Nosocomial pneumonia in the intensive care unit acquired by mechanically ventilated versus nonventilated patients. Am J Respir Crit Care Med. 2010 Dec 15;182(12):1533-9. doi: 10.1164/rccm.201001-0094OC. Epub 2010 Aug 6. PMID 20693381
- [Derived] Bello G, Pennisi MA, Di Muzio F, De Pascale G, Montini L, Maviglia R, Mercurio G, Spanu T, Antonelli M. Clinical impact of pulmonary sampling site in the diagnosis of ventilator-associated pneumonia: A prospective study using bronchoscopic bronchoalveolar lavage. J Crit Care. 2016 Jun;33:151-7. doi: 10.1016/j.jcrc.2016.02.016. Epub 2016 Mar 3. PMID 26993370